CLINICAL TRIAL: NCT07213193
Title: No-Stoma Policy in Advanced Ovarian Cancer Surgery, Feasibility and Outcomes
Brief Title: No-Stoma Policy in Advanced Ovarian Cancer Surgery
Acronym: No-Stoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7620
Record Dates: First submitted 2025-06-04; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-05

CONDITIONS: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with ovarian cancer (Experimental): Patients women who underwent colon rectal resection
  Interventions: Procedure: colon-rectal resection

INTERVENTIONS:
Procedure: colon-rectal resection — The patients who underwent colon rectal resection, would be evaluated for stomia or not.

SUMMARY:
Resection of the sigmoid-rectum is a procedure frequently required in cytoreductive surgery for advanced ovarian cancer, and it is also among the procedures with the highest risk of complications. One of the major, albeit uncommon, complications of intestinal anastomosis is anastomotic leakage. According to the literature, the rate of anastomotic leakage following cytoreductive surgery for ovarian cancer ranges from 1.7% to 17%.

The risk factors associated with this complication are varied and often inconsistent across studies. They range from preoperative clinical conditions-such as age, low albumin levels, and Body Mass Index < 18-to intraoperative factors such as low to mid rectal resection, high ligation of the inferior mesenteric artery, and multiple bowel resections.

Apart from the rehabilitative programs introduced by the Enhanced Recovery After Surgery protocol-which aim to improve the nutritional status of patients undergoing cytoreductive surgery for ovarian cancer-we currently lack validated tools to reduce the risk of leakage. The most commonly used strategy remains the creation of a protective stoma. However, several studies have shown that this procedure is not actually a protective factor against anastomotic leakage; rather, its utility lies in mitigating the severity of the complication.

Nonetheless, stomas have a significant clinical and psychological impact, with complication rates ranging from 33.9% to 45% and reversal rates between 66.5% and 89%.

This study aims to evaluate the feasibility of a no-stoma strategy in a selected "low-risk" population for anastomotic leakage among patients undergoing cytoreductive surgery for primary or recurrent ovarian cancer. Focusing on the goal of achieving a zero stoma rate, the study will provide valuable insights into the utility and outcomes of stoma creation. The results will support more informed and patient-centered clinical decisions in the management of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or anatomopathological diagnosis of malignant ovarian tumor undergoing elective primary or secondary cytoreduction and needing rectosigmoid resection and anastomosis
* Informed consent signed prior to performing any procedure related to the clinical trial
* Age 18 years old.

Exclusion Criteria:

* Patients with histologies other than ovarian tumor.
* Only palliative surgery planned
* Patients who do not require sigmoid-rectum resection after intraoperative evaluation
* Patients who do not receive colorectal anastomosis and undergo end ostomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Anastomotic Dehiscence in Low-Risk Patients Undergoing Primary or Secondary Cytoreductive Surgery for Ovarian, Fallopian Tube, or Peritoneal Tumors | Intraoperative and postoperative follow-up period (90 days postoperative)
  The feasibility of a no-stoma policy will be assessed by calculating the rate of anastomotic dehiscence in low-risk patients (who therefore did not receive a diverting stoma) and comparing these results with published data from the literature.

SECONDARY OUTCOMES:
Risk Factors for Anastomotic Leak | preoperative, intraoperative
  Identification of preoperative and intraoperative variables associated with anastomotic leak using a multivariable logistic regression model.
Rate of Occult Anastomotic Leak in Patients With Diverting Ostomy | Postoperative days up to 20.
  Proportion of asymptomatic patients with diverting ostomy presenting with occult anastomotic leak, as assessed by water-soluble rectal contrast enema performed between postoperative days 5 and 10.
Management Strategies for Anastomotic Leak | Postoperative period (up to 90 days).
  Description and distribution of management strategies for anastomotic leak (conservative vs. non-conservative), stratified by low- and high-risk patient groups, and evaluation of the role of ostomy in leak management.
Impact of Bowel Surgery on Quality of Life | Baseline (pre-surgery), 3 months, and 6 months post-surgery.
  Change in quality of life and bowel function, as measured by:
  Gastrointestinal Quality of Life Index (GIQLI) in all patients STOMA questionnaire in patients with diverting ostomy Low Anterior Resection Syndrome (LARS) score Knowles-Eccersley-Scott-Symptom (KESS) questionnaire All questionnaires will be administered preoperatively and at 3 and 6 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Vargiu, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Ginecologia Oncologica, Roma, Italy